CLINICAL TRIAL: NCT05927220
Title: WORST PATTERN OF INVASION IN ORAL SQUAMOUS CELL CARCINOMA: AN INDEPENDENT PROGNOSTIC INDICATOR
Brief Title: WORST PATTERN OF INVASION IN ORAL SQUAMOUS CELL CARCINOMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Armed Forces Institute of Pathology Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Manahil Rahat, M.Phil. Trainee in Oral and Maxillofacial Pathology, Principal Investigator, Armed Forces Institute of Pathology Rawalpindi
Other Study IDs: NUMS/AFPG/22/MPHIL/029
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Oral Cancer; Oral Cavity Cancer; Oral Squamous Cell Carcinoma
Keywords: prognosis; TNM staging; Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cohesive (I-III) worst patterns of invasion at tumor host interface
  Interventions: Diagnostic Test: Biopsy Specimens Histopathology
- non-cohesive (IV-V) worst patterns of invasion at tumor host interface
  Interventions: Diagnostic Test: Biopsy Specimens Histopathology

INTERVENTIONS:
Diagnostic Test: Biopsy Specimens Histopathology — paraffin-embedded blocks with sections from the tumor will be selected. Patterns of invasion will be recorded by for all cases by histopathologists

SUMMARY:
Cancer of the oral mucosa, also known as oral squamous cell carcinoma (OSCC), occurs as an ulceroproliferative lesion that can develop at any site in the mouth, from the lips to oropharynx. OSCC (Oral squamous cell carcinoma) is a biologically aggressive tumor and this has piqued interest in research into several prognostic histopathological indicators during the past few decades. The AJCC 8th edition TNM staging system incorporates histopathological factors including depth of invasion (DOI) that affect patient outcomes. Numerous studies have linked a poor prognosis and increased locoregional failure with certain "patterns of invasion" (POI) in OSCC. However, this factor is not utilized for treatment decision making and for outcome assessment.

The management and prognosis of oral squamous cell carcinoma (OSCC) depends on tumor stage, differentiation, perineural and lymphovascular invasion, depth of invasion, margin status, lymph node (LN) metastasis and extranodal extension. We will evaluate the relationship of these histopathological parameters with cohesive and non cohesive worst patterns of invasion (WPOI) in OSCC. The purpose of this cross-sectional study is to determine that presence of non-cohesive WPOI is associated with advanced T stage, poor differentiation, PNI, greater depth of invasion, and higher chances of nodal metastasis. WPOI is associated with poor DFS (disease free survival), treatment intensification in early stage disease with non-cohesive WPOI may improve survival.

Therefore, it should also be included in routine reporting protocol for OSCC to aid in describing the aggressive behaviour of disease.

DETAILED DESCRIPTION:
Oral cancer is one of the most often diagnosed types of the disease in Pakistan (Globocan, 2020 Pakistan). Squamous cell carcinomas account for over 90% of oral cancers (Anwar et al., 2020) . Several indicators point to a poor prognosis for OSCC, such as advanced tumor stage, higher tumor grade, extra capsular extension, nodal metastases, greater depth of invasion, lymphovascular invasion, poor differentiation, positive surgical margins, and perineural invasion have all been shown to be related with poor prognosis of patients with OSCC (Khan et al., 2023) . These factors have been rarely evaluated in Pakistani population.

Although there have been significant advances in the management of other types of cancer, OSCC still has few therapeutic options. The overall five-year survival rate for this illness remains about 50% despite substantial study over the preceding few decades.

(Chen et al., 2018) . Surgery followed by adjuvant radiation therapy and/or chemotherapy is still considered the gold standard for treating cancer. Early stage oral tongue carcinomas that are 4 mm or deeper at diagnosis, or that have a development pattern of small cell islands or satellites, should be treated as high-risk tumors requiring a multimodal approach (Lakhera et al., 2023) . Previous research into the significance of tumor budding in oral cavity malignancies has linked it to increased rates of lymph node metastases, relapse, and poor overall survival.

(Almangush et al., 2018) .Similar is seen with tumours that have greater depth of invasion. (Moeckelmann N, 2018)

The invasive tumor front is the transition zone between the tumors and the surrounding stroma. The infiltration pattern of tumors at the tumor front has been studied in a few prior investigations. (Chatterjee et al., 2019) This needs separate attention now as The College of American Pathologists now includes the reporting of oral cavity cancers based on the patterns of tumor invasion but they are not well-established prognostic variables.

(Seethala et al., 2021) This is due to the dearth of published research on the topic of invasive tumors. (Arora et al., 2017) . Despite its low prognostic value, the World Health

7

Organization's (WHO) 4th edition (2017) classification of OSCC still endorses a simple, differentiation-based histopathologic grading system that disregards important variables like tumour growth pattern and dissociation, stromal reactions (desmoplasia, local immune response), and tumor-stroma ratio. (Almangush et al., 2020) Several histological markers, easily evaluated on regular hematoxylin and eosin-stained sections, predict the outcome of OSCC. The aforementioned metrics are excellent predictors of future outcomes. These, along with WPOI, are simple and reliable prognostic indicators in early-stage OSCC that are linked to a worse prognosis. Since WPOI may aid in the individualised management of OSCC patients, it is recommended that it be evaluated in both resection and preoperative biopsy specimens as part of a standardised reporting format. (Chatterjee et al., 2019)

ELIGIBILITY:
Inclusion Criteria:

* All OSCC patients who underwent neck dissections
* Patients from all age groups and both genders

Exclusion Criteria:

* All specimens with poor fixation
* All specimens of patients having received chemotherapy and/or radiotherapy prior to the surgery
* Patients not consenting to be the part of study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the recent biopsy specimens of OSCC with neck dissection submitted to AFIP will be selected through convenience sampling method.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2023-07-03 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of Different Histopathological Factors & Patterns of Invasion | 03 months
  Correlation with cohesive (I-III) and non-cohesive (IV-V) worst patterns of invasive at tumor host interface in OSCC

CONTACTS AND LOCATIONS:
Overall Officials: Manahil Rahat, BDS, Principal Investigator — AFIP Rawalpindi Pakistan
Locations (1):
- Armed Forces Institute of Pathology, Rawalpindi, Punjab Province, Pakistan

REFERENCES:
- [Result] Chatterjee D, Bansal V, Malik V, Bhagat R, Punia RS, Handa U, Gupta A, Dass A. Tumor Budding and Worse Pattern of Invasion Can Predict Nodal Metastasis in Oral Cancers and Associated With Poor Survival in Early-Stage Tumors. Ear Nose Throat J. 2019 Aug;98(7):E112-E119. doi: 10.1177/0145561319848669. Epub 2019 May 9. PMID 31072197
- [Result] Mishra A, Das A, Dhal I, Shankar R, Bhavya BM, Singh N, Tripathi P, Daga D, Rai A, Gupta M, Sahu GC. Worst pattern of invasion in oral squamous cell carcinoma is an independent prognostic factor. J Oral Biol Craniofac Res. 2022 Nov-Dec;12(6):771-776. doi: 10.1016/j.jobcr.2022.08.027. Epub 2022 Sep 8. PMID 36159069
- See also: Globocan Cancer Observatory 2020 — https://gco.iarc.fr/
- See also: Oral cancer: Clinicopathological features and associated risk factors in a high risk population presenting to a major tertiary care center in Pakistan — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0236359